CLINICAL TRIAL: NCT06411821
Title: Phase 2 Trial of Ulixertinib for Patients With Histiocytic Neoplasms
Brief Title: Ulixertinib in People With Histiocytic Neoplasms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-282
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Histiocytic Neoplasms
Keywords: Ulixertinib (BVD-523); 23-282; Mitogen-activated protein kinase
MeSH Terms: interventions — ulixertinib

STUDY DESIGN:
Intervention Model Description: Multicenter phase 2 trial evaluating the efficacy and safety of monotherapy ulixertinib, an oral selective extracellular signalregulated kinase (ERK) inhibitor, for patients with histiocytic neoplasms:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mitogen-activated protein kinase (MAPK) pathway mutation (primary cohort) (Experimental): Patients in this study will receive ulixertinib, starting at 300 mg twice daily, for every 28-day cycle.
  Interventions: Drug: Ulixertinib
- No Mitogen-activated protein kinase (MAPK) pathway mutation identified (exploratory cohort) (Experimental): Patients in this study will receive ulixertinib, starting at 300 mg twice daily, for every 28-day cycle.
  Interventions: Drug: Ulixertinib

INTERVENTIONS:
Drug: Ulixertinib — 300 mg twice daily, for every 28-day cycle.
  Other Names: BVD-523

SUMMARY:
The researchers are doing this study is to find out whether ulixertinib is an effective and safe treatment for people with histiocytic neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed histiocytic neoplasm or histologic findings consistent with histiocytic neoplasm with confirmatory radiologic or molecular findings. Pathologic examination can be performed at any of the enrolling institutions. This qualification is made because it is well known that biopsies of histiocytic neoplasms are variable and do not always demonstrate "typical" morphologic appearance with all of the classically described elements. As a result, histiocytic neoplasms are not exclusively pathologic diagnoses-rather, they are interpretations of histologic findings in a clinical and radiologic context. These criteria were applied in NCT02649972 and will be applied in this trial
* Identified mutation in MAPK pathway genes, including but not limited to ARAF, BRAF, RAF1, NRAS, KRAS, MAP2K1, MAP2K2, and NF1 (for primary cohort; no mutation needed for exploratory cohort). Tumor mutation may be identified by tumor sequencing or cfDNA-based sequencing. Concordance between cfDNA and tumor sequencing for BRAFV600E and non-BRAF mutations in histiocytic neoplasms has been documented by our group and others
* Measurable disease according to PRC, confirmed by an investigator radiologist
* Age (a) ≥18 years prior to interim safety and efficacy analyses or (b) ≥12 years following the interim safety and efficacy analyses
* The histiocytic neoplasm must be (a) disease that is recurrent/refractory/persistent despite local therapies, chemotherapy, immunosuppression, or BRAF/MEK inhibitors OR (b) multisystem disease OR (c) single-system disease that is causing end-organ dysfunction and is unlikely to benefit from local or conventional (chemotherapy or immunosuppressive) therapies on the basis of evidence-based guidelines (e.g. symptomatic neurologic-only LCH)
* Prior treatment (chemotherapy, immunosuppression, BRAF inhibitor, or MEK inhibitor) is required and the patient must have (a) progressive disease or persistent disease (i.e. having disease measurable by PRC) or (b) intolerance or contraindication to chemotherapy, immunosuppression, BRAF inhibition, or MEK inhibition.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 (age ≥ 16) or Lansky 50-100 (age 12-15)
* Adequate renal function (according to the Cockcroft-Gault equation; creatinine ≤1.5 times upper limit of normal [ULN] or a glomerular filtration rate of ≥50 mL/min)

  * Pediatric patients (<18 years old) must have a creatinine clearance or radioisotope GFR ≥ 70 mL/min/1.73 m^2 or serum creatinine based on age/gender as follows:
  * < 13 years- 1.2 (Male),1.2 (Female)
  * 13 to < 16 years- 1.5 (Male), 1.4 (Female)

    °≥ 16 years- 1.7 (Male), 1.4 (Female)
  * The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the CDC.
  * Patients with renal impairment deemed the direct result of disease and therefore amenable to improvement with Ulixertinib treatment may be enrolled at the discretion of the treating investigator
* Adequate hepatic function (total bilirubin ≤1.5 times ULN, aspartate transaminase [AST] and- alanine transaminase [ALT] ≤3 times ULN or ≤5 times ULN if attributable to liver involvement by tumor). Patients with hepatic impairment deemed the direct result of disease and therefore amenable to improvement with Ulixertinib treatment may be enrolled at the discretion of the treating investigator.
* Adequate bone marrow function (hemoglobin ≥9.0 g/dL, platelets ≥100 x 10^9 cells/L, absolute neutrophil count ≥1.5 x 10^9 cells/L). Patients with cytopenias deemed the direct result of disease and therefore amenable to improvement with Ulixertinib treatment may be enrolled at the discretion of the treating investigator.
* Adequate cardiac function

  * Left ventricular ejection fraction >50% as assessed by multi-gated acquisition or ultrasound or echocardiography and
  * Corrected QT interval (QTc) <480 ms according to the Fridericia method (QTcF)
* Contraception

  * For women: a negative pregnancy test for those of child-bearing potential, must be surgically sterile, postmenopausal (no menstrual cycle for at least 12 consecutive months), or compliant with a medically approved contraceptive regimen during and for 3 months after the treatment period
  * For men: must be surgically sterile or compliant with a medically approved contraceptive regimen during and for 3 months after the treatment period
  * For patients aged <18 years who are not sexually active: abstinence is an acceptable form of contraception. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.
* Willing and able to participate in the trial and comply with all trial requirements
* Patients with a prior or concurrent malignancy whose natural history or treatment

  * does not have the potential to interfere with the safety or efficacy assessment of
  * the investigational agent may be included at the discretion of the site PI

Exclusion Criteria:

* Uncontrolled or severe intercurrent medical condition
* Receipt of any histiocytic neoplasm-directed therapy (chemotherapy, targeted therapy, biologic) within 28 days or 5 half-lives (whichever is shorter) before the first dose of ulixertinib. Patients previously treated with radiotherapy must have recovered from acute toxicities associated with such treatment
* Histiocytic neoplasm mandated for observation-only or first-line local therapy per established guidelines. Examples would include asymptomatic nodal RDD, asymptomatic osseous ECD, or limited cutaneous LCH
* Major surgery within 4 weeks of the first dose of ulixertinib
* Pregnant, lactating, or breast-feeding (for women)
* Any evidence of serious active infections. Patients are allowed to enroll if they have been fever free for at least 48 h
* History or current evidence of risk of retinal vein occlusion or central serous retinopathy. Examples of risk factors to be considered would include uncontrolled ocular hypertension or history of hyperviscosity.
* Concurrent therapy with drugs known to be strong inhibitors or inducers of CYP1A2, CYP2D6, and CYP3A4
* Concurrent therapy with p-glycoprotein inhibitors and sensitive substrates of CYP1A2, CYP2B6, CYP2C8, and CYP3A4/5 with narrow therapeutic indices
* Inability to swallow oral medications
* Prior stomach or duodenal resection that, in the opinion of the site PI, would affect the breakdown and absorption of the study medications. Patients with a feeding tube will also be excluded, as ulixertinib tablets cannot be taken broken, cracked or otherwise not intact. Note: ulixertinib is primarily absorbed in the duodenum, and therefore the potential inclusion of a patient with any prior stomach or duodenal resection should be discussed with the MSK PI
* Concurrent therapy with any investigational agent
* Any use of an investigational drug within 28 days or 5 half-lives (whichever is shorter). In addition, any drug toxicities should have recovered to grade 1 or less before start of the trial medication

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 1 year
  Best overall response by PET is defined as the best response, according to PRC, recorded from the first day of study treatment until disease progression, recurrence, or death. Complete response Normalization of all lesions' (target and nontarget) SUV to background SUVliver (or SUVbrain for brain lesions) Partial response ≥50% decrease from baseline in sum of SUVs of all target lesions relative to SUVliver (or SUVbrain for brain lesions only) Progressive disease ≥50% increase from nadir in sum of SUV of all target lesions relative to SUVliver (or SUVbrain for brain lesions only), with a minimal absolute increase of 3 units of SUV per target lesion (e.g., SUV 3 to SUV 6) New evaluable lesions deemed to represent unequivocal disease progression* Stable disease Does not meet other criteria

CONTACTS AND LOCATIONS:
Overall Officials: Eli Diamond, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Mayo Clinic (Data Collection Only), Rochester, Minnesota
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm